CLINICAL TRIAL: NCT03471754
Title: Pilot Study Using Transcranial Electrostimulation (TESA-HB) Therapy for the Treatment of Depressive Symptoms Associated With Mild to Moderate Depressive Episodes
Brief Title: Pilot Study Using Transcranial Electrostimulation (TESA-HB) Therapy for the Treatment of Depressive Symptoms
Acronym: TESAHBPilot
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Administrative reasons, and did not meet sample size requirements
Sponsor: Annecto LLC (Other)
Collaborators: Holy Redeemer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TESAHB64-17
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Mild to Moderate Depression
Keywords: Depression, transcranial electronic stimulation, pilot, open label, safety, efficacy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Pilot, Open Label, single center trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment Arm A (Experimental): TESA-HB Device, Mode 3 (15mA). Treatment arm involves two 5-day treatment cycles over a 2-week period, with 2 days off between each of the 5-day cycles. The treatment period will as for two full weeks.
  Interventions: Device: TESA-HB Transcranial Electronic Stimulation Device

INTERVENTIONS:
Device: TESA-HB Transcranial Electronic Stimulation Device — Duration of treatment: 50 Minute Therapy sessions administered one time each day, for two 5-day cycles

SUMMARY:
This pilot study uses TESA-HB therapy for treatment of depressive symptoms associated with mild and moderate depression episodes. Primary objectives of this pilot study are to demonstrate the safety of TESA-HB Therapy, and to investigate the efficacy of TESA-HB Therapy for depressive symptoms.

DETAILED DESCRIPTION:
The primary indicator variable in this study is the Hamilton Depression Rating Scale (HAM-D21), and secondary efficacy outcomes will be measured using:

* Major Depression Inventory
* Montgomery - Asberg Depression Rating Scale (MADRS)
* Beck's Depression Inventory
* Beck's Anxiety Inventory
* Hamilton Anxiety Rating Scale (HAM-A)
* The Psychological General Well-Being Index (PGWB-S)

The safety endpoints include:

* Medication Usage Log
* Adverse Event Log

Study Population includes men and women who are:

* Diagnosed with a mild to moderate depressive episode
* Have no recent history of taking antidepressant or anti-anxiety medication within 3 months prior to baseline

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65 years old on enrollment
* Assessed by Evaluator with mild to moderate depressive episode, based on the MDI Rating Scale (20-24 mild; 25-29 moderate).
* Have average MDI pain rating score of > 20 or <29 during baseline
* Assessed by Evaluator to have mild to moderate depressive episode, based on the HAM-D21 Rating Scale (8-13 = mild; 14-17 moderate).
* Assessed by Evaluator to have mild to moderate depressive episode based on ICD-10 Diagnostic Guidelines 1,2
* Willing and able to visit 2 weeks ( 5 times per week) as a clinic outpatient to participate in this clinical investigation
* Willing and able to return to the clinic for evaluation during the follow up period - 2 weeks, 1 month (4 wks), 2 months (8 wks), and 3 months (12wks) following the completion of TESA-HB Therapy
* Willing to be monitored, fill out daily medication logs, and appear for all physician visits for baseline, treatment and follow-up period
* English speaking and able to understand and approve the consent form, and understand and provide answers on the Depression and Anxiety assessment form and the Psychological General Well-Being Index (PGWB-S) questionnaires

Exclusion Criteria:• MDI Rating Scale of < 20 or > 29

* High variability in baseline MDI scores (changes more than 30%)
* HAM-D21 Rating Scale of < 8 or > 17
* Assessed outside of mild to moderate depression episode range based on the ICD-10 Diagnostic Guidelines 1,2
* Recent history of taking Antidepressant or Antianxiety medication within 3 months prior to baseline
* Is pregnant, or may be pregnant, or plans to become pregnant during the study period
* Sensitivity to electrodes and/or their conductive gels or adhesives
* Break in skin integrity at the areas of electrode placement
* Currently suspected use of narcotic
* Presence of any implanted electronic device, cardiac stimulator, or pacemaker
* History of brain injury, including seizures, epilepsy, stroke, tumor of central nervous system, or hydrocephalus
* Acute brain injuries, infections or tumor of central nervous system
* History of heart attacks within 1year congestive heart failure
* Blood pressure: > 140 systolic and/or > 90 diastolic
* History of schizophrenia
* Previous experience with Cranial Electrotherapy Stimulator (CES) devices
* Failure to complete 80% of daily medication logs or complete a questionnaire and two physician assessments during baseline period
* Failed to complete 75% of follow up visits or failed to complete more than 2 treatments will be excluded in the per-protocol (PP) analysis
* Acute psychiatric disorders (other than depression, insomnia and/or anxiety)
* Use of psychoactive drugs (other than antidepressants and/or anxiety)
* These subjects will continue to be followed in the study, but will be classified in the intent-to-treat (ITT) group
* HRHS employees, in an effort to protect their privacy, as the study will be conducted in a Holy Redeemer facility. Additionally, this exclusion was decided upon to minimize the possibility of coercion or undue influence in relationship with Holy Redeemer employees.
* Illiterate persons, as the study requires completion of assessments tools in the home setting where the subject may/may not have assistance with reading and understanding the tools, study documents and proceedures as required.
* Uninsured persons, to financially protect them in the rare instance that medical care would be required as a result of the study treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HAM-D21) | Statistically significant improvement from baseline to end of study period (4 months)
  The HAM-D21 will be analyzed as a single measure result
Medication Usage Log | Statistically significant improvement from baseline to end of study period (4 months)
  Will be used in total, as a covariate in analysis of primary outcome

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | Statistically significant improvement from baseline to end of study period (4 months)
  Will be analyzed in total score
Major Depression Inventory (MDI) | Statistically significant improvement from baseline to end of study period (4 months)
  Will be analyzed in total score
The Psychological General Well-Being Index (PGWB-S) | Statistically significant improvement from baseline to end of study period (4 months)
  Will be analyzed in total score
Beck's Depression Inventory (BDI) | Statistically significant improvement from baseline to end of study period (4 months)
  Will be analyzed in total score
Beck's Anxiety Inventory (BAI) | Statistically significant improvement from baseline to end of study period (4 months)
  Will be analyzed in total score
Hamilton Anxiety Rating Scale (HAM-A) | Statistically significant improvement from baseline to end of study period (4 months)
  Will be analyzed in total score
Medication Usage Log (MUL) | Statistically significant improvement from baseline to end of study period (4 months)
  Will be analyzed in total score, with no covariate

CONTACTS AND LOCATIONS:
Overall Officials: Beth DuPree, MD, MD, Principal Investigator — Holy Redeemer Hospital; Yakov Katsnelson, MD, Study Director — Annecto LLC
Locations (1):
- Holy Redeemer Health Care at Bensalem, 3300 Tillman Drive, Bensalem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No